CLINICAL TRIAL: NCT03624868
Title: A Randomized Pilot Trial of Tai Chi Compared to Wellness Education for Older Veterans
Brief Title: Tai Chi and Wellness Education for Older Veterans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped after completing 2 cohorts instead of the intended 3 cohorts. This was due to logistical issues and budget-related issues (timing of being able to spend the funds).
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: National Institute on Aging (NIA) (NIH); Boston University (Other)
Responsible Party: Principal Investigator, Anica Pless Kaiser, Clinical Research Psychologist, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P30AG048785 (NIH); P30AG048785 (NIH)
Record Dates: First submitted 2018-08-03; First posted 2018-08-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; PTSD; Satisfaction
Keywords: Tai Chi; Older Veterans; Physical activity; PTSD
MeSH Terms: conditions — Motor Activity; Stress Disorders, Post-Traumatic; Personal Satisfaction | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to Tai Chi or Wellness Education
Who Masked: Outcomes Assessor
Masking Description: Pre- and Post-intervention assessments will be conducted by an assessor who is blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi (Experimental): A Tai Chi protocol designed for use with older veterans will be used. In each class, the instructor will explain exercise theory and procedures of Tai Chi and review printed materials. Every session will include the following components: (1) warm-up and a review of Tai Chi principles; (2) Tai Chi movement; (3) breathing techniques; (4) relaxation. Each component of the program derives from classical Yang style Tai Chi 108 posture. The Tai Chi instructor will also encourage patients to practice for at least 30 minutes a day at home and to complete daily logs indicating the amount of time that they spent engaged in Tai Chi exercise. Discussion of goal-setting regarding home practice and solutions to potential barriers will be included.
  Interventions: Behavioral: Tai Chi
- Wellness Education (Active Comparator): The wellness education intervention will correspond to the VA Whole Health Program to emphasize wellness across various domains (e.g., physical, emotional, and spiritual lives). The Whole Health program focuses on teaching mindful awareness to promote behavioral changes that are consistent with an individual's health goals. Components of the Whole Health model include working the body, surroundings, personal development, food and drink, recharge, family, friends and coworkers, spirit and soul, and power of the mind. Each session will include a video clip as well as a brief mindfulness exercise that corresponds with the material being presented. Goal-setting using the SMART goals model, with regards to health and wellness, and discussions about ways to address potential barriers will be included in this condition.
  Interventions: Behavioral: Wellness Education

INTERVENTIONS:
Behavioral: Tai Chi — See above description
  Arms: Tai Chi
Behavioral: Wellness Education — See above description
  Arms: Wellness Education

SUMMARY:
The primary purpose of this study is to examine physical fitness, PTSD, and satisfaction with a Tai Chi intervention for older (aged 60 and older), sedentary, trauma-exposed veterans, in comparison to a wellness education attention control. Secondary outcomes include physical activity, depression, well-being, late-onset stress, functional status, cognition, and exercise self-efficacy. Outcomes will be examined pre- to post-intervention and in comparison to the control condition.

DETAILED DESCRIPTION:
The proposed study will consist of a pilot trial of three 12-week, 24-session Tai Chi intervention groups compared with three 12-week, 24-session wellness education control groups. Participants will be randomly assigned in blocks of 14 to either the Tai Chi or the wellness education condition, half to each. Veterans who do not agree to randomization will be excluded. Baseline and post-intervention assessments will be completed, and it is anticipated that 42 individuals will complete baseline assessments. After the final sessions, participants will be asked to provide feedback to investigators via questionnaires, a focus group discussion, and individual interviews utilizing open-ended questions. Information collected from participants will be integrated and utilized for presentations/manuscript preparation, as well as to refine protocols for use in future research.

Potentially eligible veterans who have expressed interest in the study will be called and research staff will describe all aspects of the study. Research staff will answer any questions, and then obtain oral consent for screening for eligibility criteria in the medical record. Study staff will then go through the eligibility criteria over the telephone and schedule a baseline assessment as appropriate. Participants will be mailed information about the time and location for the initial baseline assessment and the class schedule and location to which they are assigned. They will also receive phone calls with this information. Information collected during the telephone screening (prior to completion of the Informed Consent Form) will be collected and retained with the prospective participant's verbal permission. This information will be kept separate from identifying information (names, addresses, and telephone numbers). Some information collected from the electronic medical record will be recorded in order to document inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Have experienced a traumatic event (determined through telephone screening)
* English-speaking
* Considered to be sedentary
* Not planning to relocate in the next three months
* Reports ability to attend group sessions.

Exclusion Criteria:

* Lacks the capacity to provide consent
* Unable to stand for the duration of a 60-minute Tai Chi intervention
* Has major medical, psychiatric, or neurological disorder or has a moderate or severe traumatic brain injury,
* Change in psychotropic or pain medication during the past month
* Regular current Tai Chi, formal mindfulness meditation program, or yoga practice
* Unwillingness to be randomly assigned to group
* Engagement in another treatment study that might impact findings

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test | at pre-intervention and at post-intervention, about 12 weeks
  Physical fitness
Posttraumatic Stress Disorder Checklist (PCL-5) | at pre-intervention and at post-intervention, about 12 weeks
  PTSD checklist

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | at pre-intervention and at post-intervention, about 12 weeks
  Physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Anica Pless Kaiser, PhD, Principal Investigator — VA Boston Healthcare System and Boston University School of Medicine
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No